CLINICAL TRIAL: NCT01443962
Title: The Effect of PEEP on Regional Cerebral Oxygen Saturation During Laparoscopic Cholecystectomy
Brief Title: The Effect of Positive End Expiratory Pressure (PEEP) During Laparoscopic Cholecystectomy
Acronym: lapaPEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Jeong Kwak, Associate professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GIRBA 2568
Record Dates: First submitted 2011-09-27; First posted 2011-09-30 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Brain Ischemia
Keywords: laparoscopic cholecystectomy; PEEP; rSO2
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zero positive end expiratory pressure (Experimental): Number: 30, apply no PEEP during the pneumoperitoneum during the laparoscopic cholecystectomy PEEP was not applied whole investigation period
  Interventions: Other: PEEP
- positive end expiratory pressure (Active Comparator): applying PEEP 10 cmH2O during pneumoperitoneum continuously
  Interventions: Other: ZEEP

INTERVENTIONS:
Other: PEEP — applying PEEP 0 cmH2O during pneumoperitoneum continuously
  Other Names: PEEP 0
  Arms: Zero positive end expiratory pressure
Other: ZEEP — applying PEEP 10 cmH2O during pneumoperitoneum continuously
  Other Names: PEEP 10
  Arms: positive end expiratory pressure

SUMMARY:
During the laparoscopic cholecystectomy, Pneumoperitoneum could affect to the regional oxygen saturation of brain. positive end expiratory pressure (PEEP)could improve the respiratory parameters include oxygenation. So applying PEEP could improve the regional brain oxygen saturation (rSO2)

DETAILED DESCRIPTION:
During the laparoscopic cholecystectomy, Pneumoperitoneum could affect to the regional oxygen saturation of brain due to increased intracranial pressure, central venous pressure and make worse to respiratory parameters. Positive end expiratory pressure could improve the respiratory parameters include oxygenation. So applying PEEP could improve the regional oxygen saturation of brain during the pneumoperitoneum during the laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II,
* 20-65 year,
* patient who undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* cerebrovascular disease,
* coronary artery disease,
* morbid obesity (BMI > 30)
* propofol allergy,
* addictive

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
change in regional brain oxygen saturation | from baseline record rSO2 every 10 minutes
  FiO2 0.6, Tidal vlume 8 ml/IBW (kg), PEEP 10 cm H2O or not, respiratory rate as end-tidal carbone dioxide concentration (ETCO2). During the peumoperitoneum record rSO2 every 10 minutes with respiratory parameters (Peak pressure, mean pressure, PEEP) and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Chon Lee, M.D., Ph.D, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Hyun Jeong Kwak, Incheon, South Korea